CLINICAL TRIAL: NCT03602807
Title: Safety and Effect of Low-Energy Extracorporeal Shockwave Therapy (ESWT) on the Renal Allograft in Transplant Recipients - a Pilot Study.
Brief Title: Safety and Effect of Low-Energy Extracorporeal Shockwave Therapy (ESWT) on the Renal Allograft in Transplant Recipients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Ronja Niemann Lundrup, Undergraduate researcher, BSc.med, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESWT-tx
Record Dates: First submitted 2018-06-19; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Transplant Dysfunction
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental)
  Interventions: Device: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — 2 treatments a week for 3 weeks consisting of 3000 focused shockwaves of 4Hz and 0,20mJ/mm2 applied over the kidney allograft.
  Treatment is performed using the STORZ DUOLITH® SD1 T-TOP "F-SW ultra"

SUMMARY:
The aim is to investigate the safety and potential effect of Low-energy Shockwave Therapy (ESWT) on the transplanted kidney. The treatment consist of ESWT two times a week for three weeks, six treatments in total.

The hypothesis is that ESWT with improve the renal function, by reducing proteinuria (in a 24-hour urine collection test) and improving renal clearance of 51Cr-EDTA.

The safety of ESWT on the renal allograft will be assessed during and after treatments.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 1 year ago since last kidney transplant
* P-Creatinin under 300, in the last 3 blood-samples
* U-Albumine/creatinine ratio over 100, in the last 3 urine-samples

Exclusion Criteria:

* Not Danish speaking.
* Obstructive uropathy
* Suspected autoimmune disease in the kidney graft
* Symptomatic urinal tract infection (UTI)
* Severe psychiatric disorder
* Pregnant or planning on becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in renal clearance (GFR) | At baseline and 3 months after treatment
  Comparing GFR before and 3 months after treatment sessions

SECONDARY OUTCOMES:
Change in albumin/creatine ratio in 24hour urine sample | At baseline, 1 month after treatment and 3 months after treatment
  Comparing the results from a sample of 24-hour urine sample before, 1 month after and 3 months after treatment.
Incidens of treatment-related adverse events | up to 4 months
  The participants answer questions about side-effects before and after each treatment session, at 1 month followup and 3 month followup.
  After 1 month a ultrasound of the kidney will show if there is any bleeding in the graft-tissue after the 6 treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

REFERENCES:
- [Derived] Klomjit N, Lerman A, Lerman LO. It Comes As a Shock: Kidney Repair Using Shockwave Therapy. Hypertension. 2020 Dec;76(6):1696-1703. doi: 10.1161/HYPERTENSIONAHA.120.14595. Epub 2020 Nov 2. PMID 33131308